CLINICAL TRIAL: NCT06834854
Title: Opioid Free Anesthesia in Shoulder Arthroscope
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS149/2024
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Measure Time to First Rescue Analgesia Following Extubation
MeSH Terms: interventions — Fentanyl; Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- opioid-anesthesia group (OA group)(control group) (Active Comparator)
  Interventions: Drug: fentanyl
- opioid free anesthesia group (OFA group) (Active Comparator)
  Interventions: Drug: Lidocaine (drug)

INTERVENTIONS:
Drug: fentanyl — Induction: After pre-oxygenation with 100% oxygen, anesthesia will be induced with propofol 2mg/kg (1 ampoule contains 200 mg in 20cc syringe), 100 ml of isotonic saline over 15 minutes. Fentanyl 1 mcg/kg (1 ampoule contains 100mcg over 10cc syringe). Cis-atracurium 0.2 mg/kg (1ampoule contains 20mg in 10cc syringe) will be administered and endotracheal intubation will be done
  Maintenance: Anesthesia will be maintained with Isoflurane 1-1.5 % in oxygen and air mixture 1:1, and cis-atracurium will be administered in incremental doses of 0.03mg/kg/30min. Another IV cannula will be placed with two infusion pumps of normal saline 50cc and fentanyl infusion 1-2 mcg/kg/hour (max 300 mcg total).
  Arms: opioid-anesthesia group (OA group)(control group)
Drug: Lidocaine (drug) — Induction: After pre-oxygenation with 100% oxygen, anesthesia will be induced with IV propofol 2mg/kg (1 ampoule contains 200 mg in 20cc syringe), lidocaine 2% (1.5 mg/kg (7.5cc bolus dose)), MgSO4 10% (50 mg/kg in 100 ml of isotonic saline over 15 minutes), Cis-atracurium 0.2 mg/kg (1ampoule contains 20mg in 10cc syringe) will be administered and endotracheal intubation will be done.
  Maintenance: Anesthesia will be maintained using Isoflurane 1-1.5 % in oxygen and air mixture 1:1, and cis-atracurium will be administered in incremental doses of 0.03 mg/kg/30min. Another IV cannula will be placed with 2 infusion pump one of them containing mixture of (lidocaine 2% 1.5 mg/kg/hour as infusion along with MgSO4 10% in 10-15 mg/kg/hour with 50cc normal saline over 50ml/hour), while the second contains propofol at 6-10 mg/kg/hour.
  Arms: opioid free anesthesia group (OFA group)

SUMMARY:
The investigators will assess opioid free anesthesia technique as regards effectiveness & duration of post operative analgesia in shoulder arthroscpe surgeries

DETAILED DESCRIPTION:
A. Preoperative evaluation will be done on the arrival of the patients to the theatre complex, the intravenous (IV) cannula will be introduced. Pre-loading will be done using IV crystalloids 10 mL/kg. Pre-emptive analgesia will be given using IV dexamethasone 8 mg and IV paracetamol 15 mg/kg, midazolam 2 mg, pantoprazole 40 mg and granisteron 1mg. Baseline parameters such as heart rate (HR), mean arterial pressure (MAP), oxygen saturation (SpO2) monitoring will be recorded.

Before induction of general anesthesia, Patients will be randomly assigned to opioid-free anesthesia (OFA) or opioid anesthesia (OA) (control group) using a generated randomization list.

B. intraoperative setting for both groups :

OFA group:

Induction: After pre-oxygenation with 100% oxygen, anesthesia will be induced with IV propofol 2mg/kg (1 ampoule contains 200 mg in 20cc syringe), lidocaine 2% (1.5 mg/kg (7.5cc bolus dose)), MgSO4 10% (50 mg/kg in 100 ml of isotonic saline over 15 minutes), Cis-atracurium 0.2 mg/kg (1ampoule contains 20mg in 10cc syringe) will be administered and endotracheal intubation will be done.

Maintenance: Anesthesia will be maintained using Isoflurane 1-1.5 % in oxygen and air mixture 1:1, and cis-atracurium will be administered in incremental doses of 0.03 mg/kg/30min. Another IV cannula will be placed with 2 infusion pump one of them containing mixture of (lidocaine 2% 1.5 mg/kg/hour as infusion along with MgSO4 10% in 10-15 mg/kg/hour with 50cc normal saline over 50ml/hour), while the second contains propofol at 6-10 mg/kg/hour

OA group (Control group):

Induction: After pre-oxygenation with 100% oxygen, anesthesia will be induced with propofol 2mg/kg (1 ampoule contains 200 mg in 20cc syringe), 100 ml of isotonic saline over 15 minutes. Fentanyl 1 mcg/kg (1 ampoule contains 100mcg over 10cc syringe). Cis-atracurium 0.2 mg/kg (1ampoule contains 20mg in 10cc syringe) will be administered and endotracheal intubation will be done.

Maintenance: Anesthesia will be maintained with Isoflurane 1-1.5 % in oxygen and air mixture 1:1, and cis-atracurium will be administered in incremental doses of 0.03mg/kg/30min. Another IV cannula will be placed with two infusion pumps of normal saline 50cc and fentanyl infusion 1-2 mcg/kg/hour (max 300 mcg total).

During surgery, if the patient showed hypertension (increase in MAP above 100) or tachycardia (HR above 100 beat/min) will be treated by increasing the rate of infusion

All infusions will be stopped 20 min before the end of surgery.

Recovery:

At the end of surgery, muscle relaxation will be reversed with neostigmine (0.0 5 mg/Kg) and atropine (0.02 mg/kg).

Patients will be kept after extubating for observation in PACU until fulfilling an Aldrete score of 9 Post-operative analgesia will be offered in regular doses of paracetamol 1 gm IV every 6 hours for the following 24 hours, and rescue doses of IM pethidine 25 mg (up to 100 mg max) if VAS score is >4. Total dose of rescue pethidine used will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Age group: 18-65 years old Undergoing a scheduled shoulder arthroscope

Exclusion Criteria:

Allergies to any of the study drugs. Severe bradycardia or uncontrolled hypertension preoperatively. Renal failure. Hepatic failure. Cerebral insufficiency. Pregnant or breastfeeding women. Patients' refusal to participate in the study ASA physical status class > 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Measure time to first rescue analgesia following extubation | 24 hour post-extubation

SECONDARY OUTCOMES:
Total postoperative analgesia consumption during the 24 hours following extubation | 24 hour post-extubation
Postoperative pain score for 24 hours using the Visual Analogue Scale (VAS): 30 min after recovery, hourly for 2 h and every 6 h for 24 h | 24 hour post-extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP
Access Criteria: free